CLINICAL TRIAL: NCT02334475
Title: Steroid Versus Platelet Rich Plasma in Ultrasound Guided Sacroiliac Joint Injection for Chronic Low Back Pain
Brief Title: Steroid Versus Platelet Rich Plasma Injection for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, varun singla, Dr Varun Singla, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9154/PG-2Trg/2012/20886
Record Dates: First submitted 2014-10-14; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP (P) (Experimental): Ultrasound guided sacroiliac joint injection of 3 ml of leukocyte free platelet rich plasma with 0.5 ml of calcium chloride(total volume 3.5 ml) per course. Single injection per course is being given.
  Interventions: Biological: Platelet Rich Plasma
- GROUP (S) (Active Comparator): Ultrasound guided sacroiliac joint injection of 1.5 ml of methylprednisolone (40mg/ml) and 1.5 ml of 2% lidocaine (20mg/ml) with 0.5 ml of saline (total volume 3.5 ml). Single injection per course is being given.
  Interventions: Biological: methylprednisolone

INTERVENTIONS:
Biological: Platelet Rich Plasma — single intraarticular injection of 3 ml of leukocyte free platelet rich plasma with 0.5 ml of calcium chloride(total volume 3.5 ml)
  Arms: GROUP (P)
Biological: methylprednisolone — single injection 1.5 ml of methylprednisolone (40mg/ml) and 1.5 ml of 2% lidocaine (20mg/ml) with 0.5 ml of saline (total volume 3.5 ml)
  Arms: GROUP (S)

SUMMARY:
Chronic low back pain, with or without lower extremity pain, which arises from various structures of the spine constitutes a majority of pain complaints. The sacroiliac joint (SIJ) has been implicated as the primary source of pain in 10% to 27% of patients with mechanical low back pain below L5 vertebra. The common causes of SIJ pain include a trauma like direct fall on the buttocks, a rear-end or broad-side type motor vehicle accident, and an unanticipated step into a hole or from a miscalculated height, fusion surgery, anterior dislocation, inflammatory and degenerative sacroiliac joint disease and idiopathic. The treatment of SIJ pain remains a therapeutic challenge. Besides physiotherapy and systemic therapies including non-steroidal anti-inflammatory drugs (NSAIDs) and biologic agents, intra-articular and peri articular injections of SIJ, radiofrequency neurotomy and surgical fusion are often performed for pain relief. However, the success of these interventions has been determined according to the therapeutic efficacy and correct placement of the drug. The image guidance of SIJ injections seems to be important due to the complex anatomy of the joint causing a low accuracy when performed according to clinical judgement only. The feasibility of ultrasound (USG) guided injection of SIJ has recently been demonstrated resulting in very high success rates up to 90%. Various agents being used in SIJ injections include local anaesthetics, corticosteroid, botulinum toxin-A, 12.5% dextrose, phenol-glycerine-glucose (P2G) and sodium morrhuate (cod liver oil extract). SIJ steroid injection is commonly used technique and has been found to be effective to treat SIJ pain. However, the main drawback is short term effect. Borowsky et al reported improvement in visual analog score (VAS) of 14.1% and reduction of VAS ≥ 50% in only 12.50% patients at 3 months after intra-articular steroid (2 mL 0.5% bupivacaine plus 40 mg methylprednisolone) SIJ injection. Treatment modalities being currently used do not, in general, address the disease process itself, there is clearly a need to investigate treatments that are more widely applicable for symptom management and which may also directly address the disease process itself. Current research efforts aim at modifying the rate of healing of joint by using biological healing factors which are various growth factors (transforming growth factor, vascular endothelial growth factor, fibroblast growth factor, epidermal growth factor, platelet derived growth factor etc.) found abundantly in the human blood especially in platelets. The platelet rich plasma (PRP) is an ideal autologous biological blood-derived product, which can be exogenously applied to various tissues where it releases high concentrations of platelet derived growth factors that enhance the body's natural healing response. In addition PRP possesses antimicrobial properties that may contribute to the prevention of infections. PRP is now being widely tested in different fields of medicine for its possibilities in aiding the regeneration of tissue with low healing potential. Local injection of PRP is a new modality which has been effectively used for the treatment of Achilles tendon injury in athletes, chronic epicondylar tendinopathy, chronic patellar tendinosis, rotator cuff tear, anterior cruciate ligament injury, gonoarthrosis and plantar fasciitis. The intra-articular injection of PRP into knee joint has been found to reduce the incidence of local inflammatory changes in early knee osteoarthritis. Recently, PRP has been used for low back pain caused by SIJ laxity showing significant improvement in pain scores. However, there is no study at present comparing the efficacy of intra-articular injection of PRP with corticosteroids for the treatment of chronic SIJ pain. Considering the vast potential of PRP and its safety, this study aimed at studying the efficacy of ultrasound guided intra-articular SIJ injection of leukocyte free PRP for chronic low back pain due to SIJ pathology. In the current study, we tested the hypothesis that the SIJ injection of leukocyte-free PRP may be more effective for the treatment of sacroiliac joint pain as compared with steroid injection.

ELIGIBILITY:
Inclusion criteria:

* Chronic low back pain (predominantly below L5 vertebra) of moderate intensity (visual analog scale score more than 3) for greater than 3 months
* Patients with 3 or more positive provocative tests out of 6 (Annexure-1)
* Positive X-ray, MRI or nuclear scan findings
* Failure to achieve adequate improvement with comprehensive non-operative treatments, including but not limited to activity alteration, NSAIDS, physiotherapy and/or psychological counselling

Exclusion criteria:

* Systemic infection (H/O fever, chills and/or night sweats) or localized infection at anticipated introducer entry site
* Spinal pathology that may impede recovery such as spondylolisthesis at L5/S1, or scoliosis
* Symptomatic foraminal or central canal stenosis
* H/O potentially confounding intervertebral disc disease or zygapophyseal joint pain
* Pregnancy
* Active radicular pain
* Immunosuppressive conditions (H/O TB, AIDS, cancer, diabetes, surgery <3 months)
* Allergy to medications used in the procedure
* High narcotic use (>30 mg morphine daily or equivalent)
* Contraindications pertaining to the use of platelet concentrate like history of thrombocytopenia, use of anticoagulant therapy, active infection, tumor and metastatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
pain relief as assessed by change from baseline in VAS ( VISUAL ANALOG SCALE) | 0.5, 1, 1.5 and 3 months post-intervention

SECONDARY OUTCOMES:
functional assessment using change from baseline in MODQ ( MODIFIED OSWESTRY DISABILITY QUESTIONNAIRE) | 0.5, 1, 1.5 and 3 months post-intervention
functional assessment using change from baseline in SF-12 (SHORT FORM HEALTH SURVEY) | 0.5, 1, 1.5 and 3 months post-intervention
treatment emergent adverse drug reactions | 0.5, 1, 1.5 and 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: YATINDER K BATRA, MD, Study Director — Head of Department and Professor, Anaesthesia, PGIMER, Chandigarh